CLINICAL TRIAL: NCT05289674
Title: The Effect of Lactoferrin in High Calorie Formula on IL-6 and IL10 in Children With Failure to Thrive and Infection
Acronym: Interleukin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitas Airlangga (Other)
Collaborators: Danone Institute International (Other)
Responsible Party: Principal Investigator, Andy Darma, MD, Principal Investigator on Gastroenterology, Universitas Airlangga
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: J number
Record Dates: First submitted 2022-03-05; First posted 2022-03-21 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-10

CONDITIONS: Failure to Thrive; Infections
Keywords: IL-6; High Calorie Formula; Lacoferrin; IL-10
MeSH Terms: conditions — Failure to Thrive; Infections

STUDY DESIGN:
Intervention Model Description: This study is an observational study with a pre-, post-test design
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional study with a pre-, post-test design (Experimental): After the subject are diagnosed with infection (tuberculosis/TB or urinary tract infection/ UTI), they will receive 400 kcal/day (96 g/day divided 4 times consumption) of high calorie formula prescribed by the researcher (A pediatrician) for 90 days consumption ( 8640 g). the subject will be monitored every 30 days for acceptance, tolerance, weight increment, length increment evaluation.
  The blood are withdrawn at day 0 (before invention) and day 90 (after intervention) to measure the IL-6 and IL-10 levels
  Interventions: Dietary Supplement: High Calorie Formula

INTERVENTIONS:
Dietary Supplement: High Calorie Formula — The high calorie formula is given as much as 300 kcal/day for 90 days after the subject were diagnosed with tuberculosis (TB) or urinary tract infection (UTI), determine as day 1. the diagnosis were determined by pediatrician. Before the intervention (day 0) and after the intervention (day 61), the subjects were taken the blood by laboratory employee of the private hospital in Surabaya, Indonesia

SUMMARY:
Lactoferrin is an iron-binding glycoprotein of the transferrin family which is expressed and refers to it as a "red protein from milk". It is known that lactoferrin can modulate the overall immune response in inflammatory disorders including modulation of cytokine/ chemokine production and immune regulation that resenting by interleukin (IL)-10. Children with failure to thrive have increase the risk of infectious disease. The mechanism behind this may be due to impaired of immune function, in which pro-inflammation response is increased (IL-1β, IL-6), while IL-10 acted as anti-inflammation response tends to reduces.

High calorie formula (Oral Nutrition Supplement/ONS) are products used for oral nutrition support with the aim of increasing nutritional intake. they are a nutrition treatment option for when nutrition support has been identified beside dietary counselling. ONS are typically used in addition to a normal diet, when diet alone is insufficient to meet daily nutritional requirement due to infection or others. ONS should be treated like medication, ensure they are labelled with the patient's name and provided at the prescribed time. It is well established that nutritional deficiency or inadequate can impair immune function. Growing evidence suggest that for certain nutrients increased intake above currently recommended levels may help optimize immune function including improving the defense function and thus resistance to infection while maintaining tolerance.

This study aims to analize the levels of IL-6 and IL- 10 in children with failure to thrive with infection before and after receiving the intervention of lactoferrin in high-calorie formula milk. This study is an observational study with a pre-, post-test design, with designed total subject is 80. The subject is healthy children with weight faltering aged 1-5 years diagnosed with infection (tuberculosis/TB or urinary tract infection/UTI)

DETAILED DESCRIPTION:
Interventional study with a pre-, post-test design. After the subject were diagnosed with infection (tuberculosis/TB or urinary tract infection/ UTI), they will receive 400 kcal/day (96 g/day divided 4 times consumption) of high calorie formula prescribed by the researcher (A pediatrician) for 90 days consumption (8640 g). the subject will monitored every 30 days for acceptance, tolerance, weight increment, length increment evaluation.

The blood will be withdrawn at day 0 (before invention) and day 90 (after intervention) to measure the IL-6 and IL-10 levels. The high calorie formula is given as much as 400 kcal/day for 90 days after the subject were diagnosed with tuberculosis (TB) or urinary tract infection (UTI), determine as day 1. the diagnosis will be determined by pediatrician. Before the intervention (day 0) and after the intervention (day 61), the subjects were taken the blood by laboratory employee of the private hospital in Surabaya, Indonesia

ELIGIBILITY:
Inclusion Criteria:

• Children aged 1 - 5 years were diagnosed with failure to thrive with infections (TB or UTI)

Exclusion Criteria:

* Fluid retention
* Organomegaly
* Tumor mass
* Congenital abnormalities
* Cerebral Palsy
* Hormonal disorders and syndrome

Drop out Criteria:

• Lost contact

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 75 (Actual)
Dates: Start 2021-10-04 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Acceptance and tolerance of high calorie formula by the subject | 90 days
  Change on IL-6 levels (in ng/mL), the data will be presented as mean +/- SD. The level of IL-6 will be investigated using human IL-6 ELISA kit (BT Lab)
Acceptance and tolerance of high calorie formula by the subject | 90 days
  Change on IL-10 (in ng/mL), the data will be presented as mean +/- SD. The level of IL-10 will be investigated using human IL-10 ELISA kit (BT Lab)

SECONDARY OUTCOMES:
Acceptance and tolerance of high calorie formula by the subject | 90 days
  Change on body weight (in kg) the data will be presented as mean +/- SD.The body weight will be measure using digital baby scale (Seca 354) and digital scale Seca Robusta 813.
Acceptance and tolerance of high calorie formula by the subject | 90 days
  Change on body length/body height (in cm). The body length/height will be measure using infantometer (Seca 416) and stadiometer (for children aged < 2 years, Seca 213)

CONTACTS AND LOCATIONS:
Locations (1):
- Husada Utama Hospital, Surabaya, East Java, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Widjaja NA, Hamidah A, Purnomo MT, Ardianah E. Effect of lactoferrin in oral nutrition supplement (ONS) towards IL-6 and IL-10 in failure to thrive children with infection. F1000Res. 2023 Dec 19;12:897. doi: 10.12688/f1000research.130176.3. eCollection 2023. PMID 38434639